CLINICAL TRIAL: NCT02520804
Title: Effect of Normal Saline Versus Balance Salt Solution Resuscitation on Kidney Function; A Randomized Open Label Controlled Study
Brief Title: Normal Saline Versus Balance Salt Solution Resuscitation on Kidney Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Si566/2014
Record Dates: First submitted 2015-07-29; First posted 2015-08-13 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Acute Kidney Injury; Shock
Keywords: balanced salt solution
MeSH Terms: conditions — Acute Kidney Injury; Shock | interventions — sterofundin; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal saline (Active Comparator): normal saline for fluid resuscitation and maintenance for 72 hours
  Interventions: Drug: normal saline
- sterofundin (Experimental): sterofundin for fluid resuscitation and maintenance for 72 hours
  Interventions: Drug: sterofundin

INTERVENTIONS:
Drug: sterofundin — sterofundin for shock patients in the first 72 hours
  Other Names: balance salt solution
  Arms: sterofundin
Drug: normal saline — Normal saline for shock patients in the first 72 hours
  Arms: normal saline

SUMMARY:
The purpose of this study is to determine Acute kidney injury incidence between sterofundin and normal saline ; Resuscitation shock patients

DETAILED DESCRIPTION:
Sample size:Compare proportion for independent two groups formula. n=sample size α risk of 0.05, Statistical power of 80% P1 =incidence of acute kidney injury (AKI) in control (0.6)* P2 =incidence of acute kidney injury (AKI) in balanced salt solution (0.4)** from Ratanarat R,Hantaweepant C,Tangkawattanakul N,et al.The clinical outcome of acute kidney injury in critically ill Thai patients stratified with RIFLE classification.J Med Assoc Thai 2009 Mar;92 Suppl 2:61-7.

α risk of 0.05, Statistical power of 80%

Sample size for interim analysis 1.11 x 97 = 107.67 total 108 (at least 50 cases each arm)

ELIGIBILITY:
Inclusion Criteria:

* Shock patients (hypotension with signs of poor tissue perfusion)

Exclusion Criteria:

* Age < 18 yr
* Cardiogenic shock patients (History of ST elevation and Left ventricular ejection fraction (LVEF) < 35%),
* Prolong shock >24 hrs,
* Received chloride rich crystalloid (0.9% saline) or chloride rich colloid > 1000 ml within 72 hrs before recruitment
* Do-not-resuscitation patients,
* Contraindication for IV fluid administration such as pulmonary edema.,
* Stage V chronic kidney disease (CKD),
* chronic Hemodialysis or Peritonealdialyse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | 7 day
  Number of Participants with acute kidney injury divided by KIDNEY DISEASE | IMPROVING GLOBAL OUTCOMES (KDIGO) Staging

SECONDARY OUTCOMES:
Requirement of Renal replacement therapy (RRT) | up to 7 day
sodium level | day 1-3
  change from baseline
potassium level | day 1-3
  change from baseline
chloride level | day 1-3
  change from baseline
bicarbonate level | day 1-3
  change from baseline
28-day mortality | 28 days after admission
  Number of Participants death within 28 day after admission
ICU mortality | ICU admission up to 28 day
  Number of Participants death at ICU within 28 day after admission
hospital stay | during hospital admission up to 28 day
  number of Hospital admission date
ICU hospital stay | during admission up to 28 day
  number of Hospital admission date
mean arterial pressure | day1-3
  mmHg (average)
dose of norepinephrine | day1-3
  (µg/k/min)
dose of adrenaline | day1-3
  (µg/k/min)

CONTACTS AND LOCATIONS:
Overall Officials: Ranistha Ratanarat, MD, Principal Investigator — Mahidol University
Locations (1):
- Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Barber AE, Shires GT. Cell damage after shock. New Horiz. 1996 May;4(2):161-7. PMID 8774792
- [Background] Kristensen SR. Mechanisms of cell damage and enzyme release. Dan Med Bull. 1994 Sep;41(4):423-33. PMID 7813251
- [Background] Kumar A, Parrillo J. Shock: Classification,Pathophysiology, and Approach to Management. In: Dellinger R, Parillo J,eds. Critical Care Medicine: Principles of Diagnosis and Management in the Adult. Philadelphia: Mosby Elsevier,2008.
- [Background] Marino PL.Inflammatory shock syndrome. In:Marino PL,eds. Marino's The ICU Book 4th edition.Philadelphia:Wolters Kluwer,2014.
- [Background] Myburgh JA, Mythen MG. Resuscitation fluids. N Engl J Med. 2013 Sep 26;369(13):1243-51. doi: 10.1056/NEJMra1208627. No abstract available. PMID 24066745
- [Background] Martini WZ, Cortez DS, Dubick MA. Comparisons of normal saline and lactated Ringer's resuscitation on hemodynamics, metabolic responses, and coagulation in pigs after severe hemorrhagic shock. Scand J Trauma Resusc Emerg Med. 2013 Dec 11;21:86. doi: 10.1186/1757-7241-21-86. PMID 24330733
- [Background] Chowdhury AH, Cox EF, Francis ST, Lobo DN. A randomized, controlled, double-blind crossover study on the effects of 2-L infusions of 0.9% saline and plasma-lyte(R) 148 on renal blood flow velocity and renal cortical tissue perfusion in healthy volunteers. Ann Surg. 2012 Jul;256(1):18-24. doi: 10.1097/SLA.0b013e318256be72. PMID 22580944
- [Background] Guidet B, Soni N, Della Rocca G, Kozek S, Vallet B, Annane D, James M. A balanced view of balanced solutions. Crit Care. 2010;14(5):325. doi: 10.1186/cc9230. Epub 2010 Oct 21. PMID 21067552
- [Background] Perner A, Haase N, Guttormsen AB, Tenhunen J, Klemenzson G, Aneman A, Madsen KR, Moller MH, Elkjaer JM, Poulsen LM, Bendtsen A, Winding R, Steensen M, Berezowicz P, Soe-Jensen P, Bestle M, Strand K, Wiis J, White JO, Thornberg KJ, Quist L, Nielsen J, Andersen LH, Holst LB, Thormar K, Kjaeldgaard AL, Fabritius ML, Mondrup F, Pott FC, Moller TP, Winkel P, Wetterslev J; 6S Trial Group; Scandinavian Critical Care Trials Group. Hydroxyethyl starch 130/0.42 versus Ringer's acetate in severe sepsis. N Engl J Med. 2012 Jul 12;367(2):124-34. doi: 10.1056/NEJMoa1204242. Epub 2012 Jun 27. PMID 22738085
- [Background] Ratanarat R, Hantaweepant C, Tangkawattanakul N, Permpikul C. The clinical outcome of acute kidney injury in critically ill Thai patients stratified with RIFLE classification. J Med Assoc Thai. 2009 Mar;92 Suppl 2:S61-7. PMID 19562988
- [Background] Yunos NM, Bellomo R, Hegarty C, Story D, Ho L, Bailey M. Association between a chloride-liberal vs chloride-restrictive intravenous fluid administration strategy and kidney injury in critically ill adults. JAMA. 2012 Oct 17;308(15):1566-72. doi: 10.1001/jama.2012.13356. PMID 23073953
- [Background] Shaw AD, Bagshaw SM, Goldstein SL, Scherer LA, Duan M, Schermer CR, Kellum JA. Major complications, mortality, and resource utilization after open abdominal surgery: 0.9% saline compared to Plasma-Lyte. Ann Surg. 2012 May;255(5):821-9. doi: 10.1097/SLA.0b013e31825074f5. PMID 22470070
- [Background] Kidney disease: Improving Global outcomes (KDIGO) Acute kidney injury Work Group. KDIGO Clinical Practice Guideline for Acute Kidney injury.Kidney inter., Suppl.2012;2:1-138